CLINICAL TRIAL: NCT02122289
Title: Interest of the New Technologies to Detect précocément a Respiratory Exacerbation at Patients Reached by Cystic Fibrosis.
Brief Title: Muco Smartphone Exacerbation
Acronym: MUSE
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 9172
Record Dates: First submitted 2014-04-22; First posted 2014-04-24 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Cystic Fibrosis
Keywords: Exacerbation, QoL
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Application of Smartphone (Experimental): Weekly questionnaire on Smartphone
  Interventions: Device: Application of Smartphone
- No application Smartphone (Placebo Comparator): No Weekly questionnaire on Smartphone
  Interventions: Other: No application Smartphone

INTERVENTIONS:
Device: Application of Smartphone — Weekly questionnaire on smartphone
  Arms: Application of Smartphone
Other: No application Smartphone — No weekly questionnaire on smartphone
  Arms: No application Smartphone

SUMMARY:
Exacerbation in cystic fibrosis play an important role in terms of mortality and morbidity. Exacerbation frequencies is relatedto FEV1 decline and mortality. There is a relationship between exacerbation frequency and QoLdeterioration. Moreover exacerbation treatments present health costs burden leading to important physical psychological and social impact. Preventing exacerbation and early detection of these exacerbations may decrease intensity and freqauency of exacerbation leading to increase clinical status and QoLwith a decreased health cost.

Patients actually follow in CRCM track exacerbations when visits out patient clinic and during phone call. If patients did not call or did not present regularly to out patient clinic, exacerbation detection came later and so increasde the burden and therapeutic pressure.

The objective of our study is to identify earlier the potential exacerbations and so decreased the health costs and increased the patient's QoL. Forthis purpose we propose to use modern technologiessuch as smartphone in order to create alert when patients report weekly health satatus. We will compra patients randomize in control group with standart follow-up to patients randomize in the smartphone group.Moreover we will study the compliance and satisfactory degree of the use of this device in the interventional arm.

DETAILED DESCRIPTION:
Exacerbation in cystic fibrosis play an important role in terms of mortality and morbidity. Exacerbation frequencies is relatedto FEV1 decline and mortality. There is a relationship between exacerbation frequency and QoLdeterioration. Moreover exacerbation treatments present health costs burden leading to important physical psychological and social impact. Preventing exacerbation and early detection of these exacerbations may decrease intensity and freqauency of exacerbation leading to increase clinical status and QoLwith a decreased health cost.

ELIGIBILITY:
Inclusion criteria:

* CF diagnosis
* Patient able to receive phone call
* Patient who use regulary a smartphone
* age from 14 to 25
* Patients with at least 2 exacerbations before the entry.
* Stable patient at V1

Exclusion criteria:

* Patients who are include in an interventional study
* Patient who is not able to read French language
* Patients with psychological disorder

Ages: 14 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2014-04; Primary Completion 2015-05 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Frequency of exacerbation | up to 6 months

SECONDARY OUTCOMES:
Satisfactory status and compliance | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Raphael CHIRON, Principal Investigator — University Hospital, Montpellier
Locations (2):
- France (2):
  - CRCM, Giens
  - CRCM, Montpellier